CLINICAL TRIAL: NCT03294083
Title: A Phase 1b/2a Dose-escalation and Safety/Efficacy Evaluation Study of Pexa-Vec (Thymidine Kinase-Deactivated Vaccinia Virus Plus GM-CSF) in Combination With Cemiplimab (REGN2810; Anti-PD-1) in Patients With Metastatic or Unresectable Renal Cell Carcinoma (RCC)
Brief Title: A Study of Recombinant Vaccinia Virus in Combination With Cemiplimab for Renal Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SillaJen, Inc. (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JX594-REN026
Record Dates: First submitted 2017-09-19; First posted 2017-09-26 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-08

CONDITIONS: Renal Cell Carcinoma
Keywords: Cancer; Renal cell carcinoma; Clear cell renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1, Dose escalation (Experimental): Pexa-Vec will be administered via IV infusion at a dose of 3 x 10^8 pfu once per week for 4 treatments. Based on the occurrence of dose-limiting toxicities, patients may subsequently be enrolled to receive Pexa-Vec on the same schedule at a dose of 1 x 10^9 pfu.
  Cemiplimab will be administered via IV infusion every 3 weeks.
  Interventions: Biological: Pexastimogene Devacirepvec (Pexa-Vec); Biological: Cemiplimab
- Part 2-Arm A, Pexa-Vec (IT) and Cemiplimab (Experimental): Pexa-Vec will be administered via IT (intratumoral) injection every 2 weeks for 3 treatments.
  Cemiplimab will be administered via IV infusion every 3 weeks.
  Interventions: Biological: Pexastimogene Devacirepvec (Pexa-Vec); Biological: Cemiplimab
- Part 2-Arm B, Cemiplimab (Experimental): Cemiplimab will be administered via IV infusion every 3 weeks.
  At disease progression, Pexa-Vec will be administered via IT (intratumoral) injection every 2 weeks for 3 treatments. Cemiplimab will continue every 3 weeks.
  Interventions: Biological: Pexastimogene Devacirepvec (Pexa-Vec); Biological: Cemiplimab
- Part 2-Arm C, Pexa-Vec (IV) and Cemiplimab (Experimental): Pexa-Vec will be administered via IV infusion once per week for 4 treatments.
  Cemiplimab will be administered via IV infusion every 3 weeks.
  Interventions: Biological: Pexastimogene Devacirepvec (Pexa-Vec); Biological: Cemiplimab
- Part 2-Arm D, Pexa-Vec (IV) and Cemiplimab (Experimental): Pexa-Vec will be administered via IV infusion once per week for 4 treatments.
  Cemiplimab will be administered via IV infusion every 3 weeks.
  Interventions: Biological: Pexastimogene Devacirepvec (Pexa-Vec); Biological: Cemiplimab

INTERVENTIONS:
Biological: Pexastimogene Devacirepvec (Pexa-Vec) — Pexa-Vec is a vaccinia virus based oncolytic immunotherapy designed to stimulate the immune system following infection and replication within tumor cells
  Other Names: JX-594
Biological: Cemiplimab — Cemiplimab is a monoclonal antibody to Programmed Death-1 (PD-1)

SUMMARY:
This is a Phase 1b/2a, open-label, multi-center, dose-escalation and safety/efficacy evaluation trial of Pexa-Vec plus Cemiplimab in patients with metastatic or unresectable renal cell carcinoma (RCC). The trial consists of a dose-escalation stage, where the maximum feasible dose of Pexa-Vec in combination with Cemiplimab will be determined, followed by an expansion stage. During the expansion patients will receive Cemiplimab alone or in combination with Pexa-Vec, which will be administered either through intravenous (IV) or intratumoral (IT) injection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic or unresectable clear cell renal cell carcinoma (ccRCC)
* Part 2 Arm D ONLY: Patients must be refractory to anti PD-1 or anti-PD-L1 (either as monotherapy or in-combination with other approved checkpoint inhibitors or targeted therapies according to their approved label) and patients must meet all of the following criteria:

  1. Received treatment of approved anti PD-1 or anti-PD-L1 (dosed per label of the country providing the clinical site) for at least 6 weeks. History of anti-PD-L1 only is not allowed.
  2. Progressive disease after anti PD-1 or anti-PD-L1 will be defined according to RECIST 1.1. The initial evidence of progressive disease is to be confirmed by a second assessment, no less than 4 weeks from the date of the first documented progressive disease, in the absence of rapid clinical progression. (This determination is made by the Investigator; the Sponsor will collect imaging scans for retrospective analysis. Once progressive disease is confirmed, the initial date of progressive disease documentation will be considered the date of disease progression).
  3. Documented disease progression within 12 weeks of the last dose of anti PD-1 or anti-PD-L1. Patients who were re-treated or on maintenance with anti-PD-1 or anti-PD-L1 will be allowed to enter the study as long as there is documented progressive disease within 12 weeks of the last treatment date.
* Naive to systemic therapy for RCC or have progressed after, or were intolerant of, prior systemic therapy.
* Measurable disease based on RECIST 1.1 criteria. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Karnofsky performance status of 70-100
* Age ≥20 years old (or appropriate age of consent for the region)
* Adequate hematological, hepatic, and renal function

Exclusion Criteria:

* Known significant immunodeficiency due to underlying illness (e.g., human immunodeficiency virus [HIV] / acquired immune deficiency syndrome [AIDS]) and/or immune-suppressive medication including high-dose corticosteroids
* Part 2 only: Arm A,B,C: Prior treatment with any anti-cancer immunotherapy, including therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent (prior IL-2 or interferon allowed) . For Part 1: patients are excluded if they were intolerant to anti-PD-1 or anti-PD-L1 targeted therapies
* Major surgery within 4 weeks of study treatment (minor surgical procedures are allowed)
* Ongoing severe inflammatory skin condition requiring prior medical treatment
* History of eczema requiring prior medical treatment
* Tumor(s) invading a major vascular structure (e.g., carotid artery) or other key anatomical structure (e.g., pulmonary airway) OR viable central nervous system malignancy
* Clinically significant and/or rapidly accumulating ascites, pericardial and/or pleural effusions.
* Symptomatic cardiovascular disease, including but not limited to significant coronary artery disease (e.g., requiring angioplasty or stenting) or congestive heart failure within the preceding 12 months.
* Asymptomatic cardiovascular disease (current or past history) unless cardiology consultation and clearance has been obtained for study participation.
* Inability to suspend treatment with anti-hypertensive medication for 48 hours prior to and 48 hours after all Pexa-Vec treatments
* Use of interferon/pegylated interferon (PEG-IFN) or ribavirin that cannot be discontinued within 14 days prior to any Pexa-Vec dose
* Known active Hepatitis B or Hepatitis C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose(MTD) / Maximum feasible dose (MFD) | 36 days after first treatment
  MTD/MFD of Pexa-Vec administered by IV infusion in combination with Cemiplimab
Severity and frequency of adverse events to determine safety of Pexa-Vec administered by IV infusions or IT injections in combination with IV Cemiplimab | From date of first treatment until 28 days after last treatment
  Safety will be determined by assessing the severity and frequency of adverse events and laboratory toxicity using CTCAE v4.03
Overall response rate | Every 9 weeks, then every 12 weeks after 1 year until date of first documented progression, up to 72 months
  Evaluate anti-tumor activity and efficacy of IV or IT Pexa-Vec combined with IV Cemiplimab with respect to overall response rate (ORR) per Response Evaluation Criteria In Solid Tumors (RECIST 1.1)

SECONDARY OUTCOMES:
Progression free survival | Every 9 weeks, then every 12 weeks after 1 year until date of first documented progression, up to 72 months
Disease control rate | Every 9 weeks, then every 12 weeks after 1 year until date of first documented progression, up to 72 months
Best radiographic response | Every 9 weeks, then every 12 weeks after 1 year until date of first documented progression, up to 72 months
Overall survival | Every 9 weeks, then every 12 weeks after 1 year until date of death from any cause, up to 72 months

CONTACTS AND LOCATIONS:
Locations (18):
- United States (4):
  - Site 2644 University of California, Irvine, Irvine, California
  - Site 2641 University of Miami, Miami, Florida
  - Site 2643 Washington University, St Louis, Missouri
  - Site 2646 The Ohio State University, Columbus, Ohio
- Site 2632 Flinders Medical Centre, Bedford Park, Australia
- South Korea (13):
  - Site 2612 Kyungpook National University Chilgok Hospital, Daegu
  - Site 2616 Chungnam National University Hospital, Daejeon
  - Site 2618 Chonnam National University Hwasun Hospital, Gwangju
  - Site 2622 Gachon University Gil Medical Center, Incheon
  - Site 2613 Dong-A University Hospital, Pusan
  - Site 2619 Pusan National University Hospital, Pusan
  - Site 2617 CHA University, CHA Bundang Medical Center, Seongnam
  - Site 2620 Seoul National University Bundang Hospital, Seongnam-si
  - Site 2615 Korea University Anam Hospital, Seoul
  - Site 2610 Severance Hospital, Yonsei University Health System, Seoul
  - Site 2623 Ajou University Hospital, Suwon
  - Site 2625 Wonju Severance Christian Hospital, Wŏnju
  - Site 2624 Pusan National University Yangsan Hospital, Yangsan